CLINICAL TRIAL: NCT00784498
Title: Procedural Sedation for Painful Orthopedic Manipulations With Propofol vs. Midazolam/Ketamine in the Adult Emergency Department
Brief Title: Procedural Sedation Using Propofol Versus Midazolam/Ketamine in the Adult Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Pinchas Halpern MD. Director of Department of Emergency Medicine, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-08-PH-0272-CTIL; 0272-08-TLV; Study Protocol [1] 2-Jul-08
Record Dates: First submitted 2008-11-02; First posted 2008-11-04 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2008-11

CONDITIONS: Procedural Sedation
Keywords: Procedural sedation and analgesia; Emergency Department; propofol versus ketamine and midazolam; painful orthopedic manipulations
MeSH Terms: conditions — Agnosia; Emergencies | interventions — Ketamine; Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midazolam/ketamine (Active Comparator): Patients with orthopedic injuries requiring painful manipulation
  Interventions: Drug: Ketamine/Midazolam
- propofol (Active Comparator): Patients with orthopedic injuries requiring painful manipulation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine/Midazolam — Intravenous bolus of midazolam 0.1mg/kg in titrated dose of 1 mg/min until spontaneous eye closure or up to 5mg (whichever comes first) followed by ketamine 0.5-1mg/kg (up to 100mg) in titrated dose of 10mg/30 seconds, to achieve the desired level of sedation
  Arms: midazolam/ketamine
Drug: Propofol — Intravenous bolus of propofol 0.5-1mg/kg in titrated dose of 10mg/30seconds (up to 100mg) to achieve the desired level of sedation
  Arms: propofol

SUMMARY:
The use of procedural sedation and analgesia (PSA) to accomplish painful procedures in the emergency department (ED) has become a standard of practice over the last decade. Substantial variance exists regarding usage of medication for PSA, and many anesthetic agents have been proposed for this use.

To our knowledge no head to head study compared the clinical effectiveness, safety profile and amnestic properties of midazolam/ketamine vs. propofol regimens for PSA in the adult ED setting.

This prospective randomized trail can will help to evaluate the effectiveness and safety profile of Midazolam/katamine regimen for ED PSA in adults and will contribute to the discussion regarding propofol roll in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients with orthopedic injuries requiring painful manipulation (i.e. reduction of fracture or dislocation, drainage of abscess, suture of extensive laceration)
* Age between18-65 years
* American Society of Anesthesiologists (ASA) score of 1 or 2
* Systolic blood pressure higher than 90 mmHg and lower than 160 mmHg before initiating sedation
* Willingness and ability to provide an informed consent
* No known hypersensitivity to either medication
* No evidence of intoxication
* No recent heavy meal.

Exclusion Criteria:

* Pregnant women and patients who do not meet the above criteria will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The effectiveness and safety profile of procedural sedation using propofol versus midazolam/ketamine. | outcome measures will be monitored continuously and will be documented every few minutes from initiating sedation until the patient returns to his/her basic mental status

SECONDARY OUTCOMES:
The amnestic properties of procedural sedation with propofol versus midazolam/ketamine. | Recall issues will be assessed after the patient returns to his/her basic mental status and within 72 hours from the procedure (either on a follow up visit or by a phone call)

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Halpern, MD, Principal Investigator — Tel Aviv Sourasky Medical Center, Sackler Faculty of Medicine, Tel Aviv University, Tel Aviv, Israel
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel